CLINICAL TRIAL: NCT02286297
Title: Comparison of Intubation Through the McGrath® MAC, GlideScope®, AirTraq® and Miller Laryngoscope by Paramedics During Pediatric Cardiopulmonary Resuscitation: a Randomized Crossover Manikin Trial.
Brief Title: Pediatric Endotracheal Intubation During Resuscitation
Acronym: PETI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, National Institute of Cardiology, Warsaw, Poland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ETI/2014/08
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Pediatric; Cardiopulmonary
Keywords: Intubation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endotracheal intubation without chest compressions (Experimental): Endotracheal intubation of mannikin during resuscitation without chest compressions.
  Interventions: Device: McGRATH® MAC; Device: AirTraq; Device: GlideScope; Device: Miller
- Endotracheal intubation with uninterrupted chest compressions (Experimental): Endotracheal intubation of mannikin during resuscitation with uninterrupted chest compressions. In order to simulate the difficulties associated with intubation during uninterrupted chest compressions, CPR was performed by using LUCAS-2 (Physio-Control, Redmond, WA, U.S.).
  Interventions: Device: McGRATH® MAC; Device: AirTraq; Device: GlideScope; Device: Miller

INTERVENTIONS:
Device: McGRATH® MAC — video-laryngoscopy-1
Device: AirTraq — video-laryngoscopy-2
Device: GlideScope — video-laryngoscopy-3
Device: Miller — Direct laryngoscopy

SUMMARY:
Endotracheal intubation (ETI) is perceived as the optimal method of providing and maintaining a clear and secure airway. The 2010 European Resuscitation Council (ERC) guidelines emphasized the importance of minimal interruption during cardiopulmonary resuscitation (CPR). These guidelines also suggest that skilled operators should be able to secure the airway without interrupting chest compression. The aim of the study was to compare time and success rates of different available video laryngoscopes and the Miller laryngoscope for emergency intubation during simulated pediatric CPR.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* paramedics, nurses, physicians

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2014-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Time to intubation | intraoperative
  time from insertion of the blade to the first manual ventilation of the manikin´s lungs. If time of intubation is over than 60 seconds, attempt was recognized as failure.

SECONDARY OUTCOMES:
Success of intubation | intraoperative
  effectiveness of the first, second and third intubation attempts and overall effectiveness of intubation by participants using four intubation devices. If the examinee failed at all attempts, the case was excluded from the time calculations.
Visual Analog scale (VAS) score | 1 day
  participants were asked which method they would prefer in a real-life resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — Institute of Cardiology
Locations (1):
- International Institute of Rescue Research and Education, Warsaw, Masovia, Poland